CLINICAL TRIAL: NCT07253207
Title: A Randomized, Double-Blind, Active-Controlled, Multicenter Phase III Clinical Trial Evaluating the Efficacy and Safety of Levomilnacipran Hydrochloride Extended-Release Capsules in the Treatment of Patients With Major Depressive Disorder (MDD)
Brief Title: Efficacy and Safety Study of Levomilnacipran Hydrochloride Extended-Release Capsules in Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zhejiang Huahai Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HH-ZMNPL-2024
Record Dates: First submitted 2025-11-18; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Duloxetine Hydrochloride Enteric Capsules (Active Comparator)
  Interventions: Drug: Duloxetine Hydrochloride Enteric Capsules
- Levomilnacipran Hydrochloride Extended-Release Capsules (Experimental)
  Interventions: Drug: Levomilnacipran Hydrochloride Extended-Release Capsules

INTERVENTIONS:
Drug: Levomilnacipran Hydrochloride Extended-Release Capsules — Treatment period:
  1. Levomilnacipran Hydrochloride Extended-Release Capsules 20mg/day is to be given orally, once daily, for 1-2 days in the first week of treatment.
  2. Levomilnacipran Hydrochloride Extended-Release Capsules 40mg/day is to be given orally, once daily, for 3-7 days in the first week of treatment.
  3. Levomilnacipran Hydrochloride Extended-Release Capsules 80mg/day is to be given orally, once daily, for the second week of treatment.
  4. Levomilnacipran Hydrochloride Extended-Release Capsules 40, 80 or 120mg/day (the dosage based on the participant's clinical response and tolerance) is to be given orally, once daily, for the weeks 3 to 8 of treatment.
  Reduction period: Dosage of 20-80mg/day based on the tolerable dose during the 8th week of treatment.
  Arms: Levomilnacipran Hydrochloride Extended-Release Capsules
Drug: Duloxetine Hydrochloride Enteric Capsules — Treatment period: Duloxetine Hydrochloride Enteric Capsules 60mg/day is to be given orally, once daily, for 8 weeks.
  Reduction period: Duloxetine Hydrochloride Enteric Capsules 60mg/day is to be given orally, once daily, for 2 weeks.
  Arms: Duloxetine Hydrochloride Enteric Capsules

SUMMARY:
The purpose of this study is using Duloxetine Hydrochloride Enteric Capsules as the positive control, to evaluate the efficacy and safety of Levomilnacipran Hydrochloride Extended-Release Capsules in patients with Major Depressive Disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient patients aged 18 to 65 years (inclusive of 18 but exclusive of 65), regardless of gender;
2. Meet the diagnostic criteria for depression as per the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), with a duration of at least 3 months for first-episode cases (30 days per month);
3. Current depressive episode confirmed using the Mini-International Neuropsychiatric Interview (M.I.N.I.) version 7.0.0 or higher;
4. Total HAMD17 score ≥18 at screening and baseline visits;
5. CGI-S score ≥4 at screening and baseline visits;
6. Agree to use effective contraception during the trial and for 30 days after the last dose (women of childbearing potential must have a negative pregnancy test before dosing and not be breastfeeding), and men and women must have no plans to donate sperm or eggs, respectively;
7. Voluntarily participate in the trial and sign the informed consent form.

Exclusion Criteria:

1. Meet DSM-5 diagnostic criteria for other mental disorders (including but not limited to schizophrenia spectrum and other psychotic disorders, bipolar and related disorders, obsessive-compulsive and related disorders, somatic symptom and related disorders);
2. Previous failure to respond to adequate dose and duration (maximum recommended dose for MDD as per label for at least 4 weeks) of serotonin and norepinephrine reuptake inhibitors (including but not limited to milnacipran, levomilnacipran, duloxetine, venlafaxine, desvenlafaxine), or failure to respond to adequate dose and duration of at least two antidepressant drugs;
3. Allergic to milnacipran, levomilnacipran, duloxetine, or excipients of the trial drug, or have an allergic constitution;
4. History of suicide attempt within 1 year prior to screening; suicidal or self-harming behavior during screening; HAMD17 item 3 (suicide) score ≥3; currently at high suicide risk;
5. Depression secondary to other diseases;
6. History of epileptic seizures (except for febrile convulsions in childhood);
7. Received systematic electroconvulsive therapy, transcranial magnetic stimulation, transcranial direct current stimulation, systematic psychotherapy, or other treatments with antidepressant effects within 3 months prior to screening; received electroconvulsive therapy within 1 month prior to screening;
8. Discontinuation of psychotropic drugs or their active metabolites less than 5 half-lives, or monoamine oxidase inhibitors less than 2 weeks, before randomization;
9. Required to use drugs with clinically significant interactions with the trial drug during the trial (including but not limited to monoamine oxidase inhibitors, other serotonergic drugs, drugs affecting coagulation, strong CYP3A4/CYP1A2/CYP2D6 inhibitors or inducers, alcohol, linezolid, and intravenous methylene blue);
10. Conditions affecting drug swallowing or absorption, as judged by the investigator;
11. Risk factors for angle-closure glaucoma, as judged by the investigator;
12. Abnormal and clinically significant results from physical examinations or laboratory tests at screening or baseline, as judged by the investigator, including but not limited to ALT, AST, total bilirubin, or serum creatinine >1.5 times the upper limit of normal, or thyroid-stimulating hormone outside the normal range;
13. Current or past medical history of diseases or dysfunctions affecting the trial, as judged by the investigator, including but not limited to chronic or acute diseases of the nervous, motor, circulatory, respiratory, digestive, urinary, endocrine, reproductive, or immune systems;
14. Clinically significant cardiovascular diseases, as judged by the investigator, including but not limited to atrial fibrillation, second- or third-degree atrioventricular block, myocardial infarction within 12 months, or NYHA heart function class III or above;
15. ECG QTcF interval ≥450 ms (males) or ≥470 ms (females), or other factors increasing the risk of QTcF prolongation or arrhythmic events (including but not limited to heart failure, hypokalemia, family history of long QT syndrome), or ECG heart rate <50 bpm or >120 bpm (Note: QTcF = QT/(RR^0.33));
16. Resting seated systolic blood pressure <90 mmHg or >140 mmHg, or diastolic blood pressure <50 mmHg or >90 mmHg;
17. Diagnosed with end-stage renal disease at screening or previously, as judged by the investigator;
18. History of malignant tumors, as judged by the investigator at screening or previously;
19. Positive virological screening for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb), syphilis antibody, or human immunodeficiency virus (HIV) antibody during screening;
20. History of drug or alcohol abuse;
21. Weekly alcohol consumption exceeding 14 units in the 6 months prior to screening (1 unit = 360 mL beer, 45 mL 40% liquor, or 150 mL wine);
22. Inability to comply with medication instructions, as judged by the investigator;
23. Physiological or psychological conditions that may increase trial risks, affect protocol compliance, or prevent trial completion, as judged by the investigator;
24. Participation in any clinical trial (received investigational drugs or medical devices) within 30 days before signing the informed consent form;
25. Concomitant diseases that may interfere with trial procedures or assessments, or other conditions deemed unsuitable for trial participation by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
The change from baseline in the total score of the 17-item Hamilton Depression Rating Scale (HAM-D17) after 8 weeks of treatment. | 8 weeks of treatment
  Change from baseline at Week 8 in total score of the 17-item Hamilton Depression Rating Scale (HAM-D17) (Score range: 0-52; a higher score indicates greater severity of depressive symptoms.)

CONTACTS AND LOCATIONS:
Locations (28):
- China (28):
  - Hefei Fourth People's Hospital, Hefei, Anhui
  - Wuhu Hospital of Beijing Anding Hospital, Capital Medical University, Wuhu, Anhui
  - Beijing Anding Hospital Capital Medical University, Beijing, Beijing Municipality
  - Beijing HuiLongGuan Hospital, Beijing, Beijing Municipality
  - Chongqing Mental Health Center, Chongqing, Chongqing Municipality
  - Affiliated Brain Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Hebei Provincial Mental Health Center, Baoding, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Hunan Provincial Second People's Hospital, Changsha, Hunan
  - Nantong Mental Health Center, Nantong, Jiangsu
  - Suzhou Guangji Hospital, Suzhou, Jiangsu
  - Wuxi Mental Health Center, Wuxi, Jiangsu
  - Zhenjiang Mental Health Center, Zhenjiang, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jiangxi Provincial Psychiatric Hospital, Nanchang, Jiangxi
  - Jilin Provincial Neuropsychiatric Hospital, Siping, Jilin
  - The First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi
  - Xi 'an Mental Health Center, Xi'an, Shaanxi
  - Shandong Provincial Mental Health Center, Jinan, Shandong
  - Shanghai Pudong New Area Mental Health Center, Shanghai, Shanghai Municipality
  - Linfen Central Hospital, Linfen, Shanxi
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Chengdu Fourth People's Hospital, Chengdu, Sichuan
  - Tianjin Fourth Central Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Hangzhou Seventh People's Hospital, Hangzhou, Zhejiang
  - Huzhou Third People's Hospital, Huzhou, Zhejiang
  - Ningbo University Affiliated Kangning Hospital, Ningbo, Zhejiang